CLINICAL TRIAL: NCT06422247
Title: Observational Study in Japanese Patients With Peripheral T-Cell Lymphoma Who Received Second-Line Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA073-1019
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsed or refractory peripheral T-cell lymphoma initiating second-line systemic therapy
  Interventions: Drug: Systemic therapy

INTERVENTIONS:
Drug: Systemic therapy — Approved peripheral T-cell lymphoma systemic treatments prescribed by the treating physician

SUMMARY:
The purpose of this study is to describe the therapeutic practices and the prognosis of patients with relapsed or refractory peripheral T-cell lymphoma in Japan

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with a confirmed diagnosis of the specific subtypes of peripheral T-cell lymphoma (PTCL) according to The World Health Organization (WHO) classification of lymphoid neoplasm, 4th edition defined by WHO and International Agency for Research on Cancer (IARC).
* Participates aged ≥18 years of age at diagnosis of PTCL.
* Participates who have been treated with a systemic therapy for PTCL and have initiated a systemic therapy as a second-line therapy for relapsed or refractory PTCL between April 1, 2018 and March 31, 2023.

Exclusion Criteria:

* Participates who have medical history of peripheral T-cell lymphoma (PTCL) treatment by unapproved drug in Japan as of 31 March 2024 or off-label drug for PTCL in Japan as of 31 March 2024.
* Participates who have medical history of participation to a separately defined registration study for regulatory approval in PTCL.
* Participates who have medical history of PTCL treatment in a separately defined clinical study with intervention by on-label regimen for PTCL.
* Participates judged to be inappropriate for enrollment in this study by the site investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with peripheral T-cell lymphoma in Japan initiating second-line systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From baseline until date of death from any cause or last known alive date, assessed up to 6 years

SECONDARY OUTCOMES:
Participant baseline demographics | Baseline
Participant baseline clinical characteristics | Baseline
Participant treatment sequence from initial diagnosis | From date of initial diagnosis until death from any cause or last known alive date, assessed up to 6 years
Frequency of treatment regimen by treatment line | End date of each treatment-line of therapy, assessed up to 6 years
Time to next treatment line or death (TTNT) | From date of first-line therapy initiation until death from any cause or last known alive date, assessed up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mebix, Inc, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts